CLINICAL TRIAL: NCT04186052
Title: Clinical Study Protocol for Targeting BCMA Autochimeric Antigen Receptor T Cell Infusion One-arm, Single-center, Open-label Clinical Trial of BCMA Autologous Chimeric Antigen Receptor T Cell Infusion in Patients With BCMA-positive Relapsed/Refractory Multiple Myeloma
Brief Title: Clinical Trial of BCMA CAR T Cell Infusion in Patients With BCMA-positive r/r Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Second Affiliated Hospital of Suzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-BCMA-001
Record Dates: First submitted 2019-11-05; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CAR-T cells Infusion (Experimental)
  Interventions: Biological: BCMA-CART cells

INTERVENTIONS:
Biological: BCMA-CART cells — Target BCMA chimeric antigen receptor T cell infusion

SUMMARY:
Multiple myeloma is a kind of hematological malignancy caused by the proliferation of malignant clonal plasma cells. In recent years, the emergence of new therapeutic drugs such as bortezomib and lenalidomide has significantly improved the therapeutic effect of mm. However, due to the presence of myeloma stem cells, most patients will inevitably relapse and die. With the development of biomedicine and immunology, immunotherapy with chimeric antigen receptor modified T cells has attracted great attention for its amazing efficacy. CAR-T cells carry receptors that can specifically recognize myeloma associated antigens, and their killing effect is not limited by MHC molecules. B-cell mature antigen is only expressed on the surface of B cells in germinal center, malignant and normal plasma cells, not on other normal human tissues and CD34 + hematopoietic stem cells. It is a relatively specific high expression on the surface of myeloma cells, which is an ideal target for MM immunotherapy. The aim of this study was to investigate the efficacy and safety of BCMA targeted T cell infusion in the treatment of BCMA positive multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* 1、 Chinese subjects aged 18-75
* 2、 According to the IMWG diagnostic criteria, the initial diagnosis of multiple myeloma
* 3、 The presence of measurable lesions at screening was determined by any of the following criteria：M-protein quantities≥1.0 g/dL or ≥200mg/24 hours urine collection ; Pathologically confirmed plasmacytoma; Abnormality of free light chain of serum κ / γ
* 4、 Received at least 3 lines of multiple myeloma treatment: each line has at least 1 complete treatment cycle, unless the best response to the treatment plan is recorded as Pd (according to the IMWG standard)
* 5、 Accepted a PI and an IMID
* 6、 Disease progression confirmed by examination data during or after the recent anti-myeloma treatment
* 7、 ECOG score 0 or 1
* 8、 The clinical laboratory values during the screening period meet the following criteria: Hemoglobin ≥ 8.0 g / dL (no RBC infused within 7 days before laboratory testing ); Recombinant human erythropoietin; Platelet ≥ 50 × 109 / L(There must be no blood transfusion within 7 days before the test); ANC≥0.75×109/L (Growth factor support is allowed, but support therapy must not be received within 7 days of laboratory testing) ; AST and ALT≤3.0×ULN; Total bilirubin≤2.0×ULN, except for subjects with congenital bilirubinemia, such as Gilbert syndrome (in this case, direct bilirubin ≤1.5×ULN); Corrected serum calcium ≤12.5 mg/dL（≤3.1 mmol/L） or free ionic calcium≤6.5 mg/dL（≤1.6 mmol/L）
* 9、 The high sensitivity serum pregnancy test (β - hCG) must be negative for fertile women at screening and before the first treatment with cyclophosphamide and fludarabine
* 10、 The following requirements must be observed by women with fertility: must agree to use an effective contraceptive method (annual failure rate of continuous and correct use is less than 1%), and agree to use an effective contraceptive method continuously for at least 100 days from signing the informed consent form (ICF) to receiving lcar-b38m cell preparation infusion. Effective contraceptive methods include: Non user dependent methods: 1) Implantable progestin contraceptives that inhibit ovulation; 2)IUD; 3) Vasectomy of sexual partner; User dependency method: 1) Compound hormone contraceptives (including estrogen and progesterone) that can inhibit ovulation; 2) A progestin contraceptive (oral or injectable) that inhibits ovulation
* 11、 In addition to effective contraceptive methods, male subjects must: At least 100 days after signing ICF and receiving lcar-b38m cell infusion, when having sex with fertile women, barrier contraceptive method must be agreed; Condom must be used when having sex with pregnant women; Women and men must agree not to donate eggs (eggs, oocytes) or sperm within 100 days of the study and within 100 days of receiving the cell preparation.
* 12、 Subjects must sign the ICF to demonstrate that they understand the purpose and procedures of the study and are willing to participate in the study. Informed consent must be obtained prior to the initiation of any examination or procedure that is relevant to the subject's disease standard treatment
* 13、 Willing and able to comply with the taboos and restrictions of this program

Exclusion Criteria:

* 1、 Have received CAR-T treatment targeting any target
* 2、 Have received any treatment for targeting BCMA
* 3、 Other invasive malignancies other than multiple myeloma have been diagnosed or treated, except in the following cases: malignant tumors that have undergone radical treatment, and no known active disease within ≥3 years before enrollment; or Well-treated non-melanoma skin cancer, no evidence of disease
* 4、 Previously received the following anti-tumor treatment (before the blood of the apheresis component): targeted therapy, epigenetic therapy or experimental drug therapy within 14 days or at least 5 half-lives (whichever is shorter), or Invasive experimental medical devices have been used. Monoclonal antibodies were used to treat multiple myeloma within 21 days. Receive cytotoxic treatment within 14 days. Proteasome inhibitor treatment was received within 14 days. Received immunomodulator treatment within 7 days. Received radiation therapy within 14 days. However, if the field covers ≤5% of the bone marrow reserve, the subject is eligible to participate in the study regardless of the date of the end of radiotherapy.
* 5、 In addition to alopecia or peripheral neuropathy, the toxicity of previous anti-tumor treatments must be improved to baseline levels or ≤1
* 6、 The following heart conditions occurred: New York Heart Association (NYHA) stage III or stage IV congestive heart failure; myocardial infarction or coronary artery bypass graft (CABG) before or 6 months prior to enrollment; clinically meaningful ventricular Arrhythmia, or history of unexplained syncope, non-vascular vagal or not due to dehydration; history of severe nonischemic cardiomyopathy; assessed by echocardiography or multi-circuit detection (MUGA) scan (in front of apheresis ≤ 8 weeks), impaired cardiac function (LVEF <45%)
* 7、 Systemic corticosteroid treatment at doses greater than 5 mg/day of prednisone (or equivalent dose of other corticosteroids) within 2 weeks prior to apheresis
* 8、 Received any of the following treatments: for the treatment of multiple myeloma, allogeneic stem cell transplantation. Apheresis has been tested for autologous stem cell transplantation within ≤12 weeks before blood collection
* 9、 A stroke or seizure occurred within 6 months prior to the signing of the ICF
* 10、 Screening for plasma cell leukemia (according to standard classification, plasma cells >2.0×109/L), Waldenstrom's macroglobulinemia, POEMS syndrome (multiple neuropathy, organ enlargement, endocrine disease, monoclonal protein disease) And skin changes) or primary AL amyloidosis
* 11、 Human immunodeficiency virus (HIV) seropositive
* 12、 Live attenuated live vaccine within 4 weeks before single blood collection
* 13、 Hepatitis B infection as defined by the American Society of Clinical Oncology (ASCO) guidelines. If the infection status is unknown, the infection level needs to be determined by the quantitative level.
* 14、 Hepatitis C (anti-hepatitis C virus [HCV] antibody positive or HCV-RNA quantitative test results positive) or known to have a history of hepatitis C
* 15、 Need oxygen to maintain adequate oxygen saturation
* 16、 It is known to have life-threatening allergic reactions, hypersensitivity reactions or intolerance to LCAR-B38M cell preparations or their excipients (including DMSO) (see the investigator's manual)
* 17、 Severe underlying conditions, such as evidence of a serious active virus, bacterial infection, or uncontrolled systemic fungal infection; active autoimmune disease or a history of autoimmune disease within 3 years; significant clinical evidence of dementia Mental state change
* 18、 Not conducive to the subject receiving or tolerating planned treatment at the research center, understanding any questions of informed consent, or any researcher believes that participating in the study does not meet the best interests of the subject (eg, impairing health), or any Prevent, limit or confuse the status of the assessment provided by the research programme
* 19、 Female subjects who were pregnant, breast-feeding, or planning to become pregnant during the study period or within 100 days of receiving the study treatment
* 20、 Male subjects who have a birth plan during the study period or within 100 days of receiving the study treatment
* 21、 Major surgery was performed within 2 weeks prior to apheresis, or planned to be performed during the study or within 2 weeks of the study treatment. (Note: Subjects scheduled for local anesthesia can participate in this study.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
safety(Incidence of AE or SAE of ≥ grade 3 ) | 12 weeks after infusion of the study drug
  Incidence of AE or SAE of ≥ grade 3 (refer to CTCAE version 4.03) related to the study drug within 12 weeks after infusion of the study drug

SECONDARY OUTCOMES:
Effectiveness | 12 weeks after infusion of the study drug
  ORR at 12 weeks after infusion (ORR12)

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Department of the Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided